CLINICAL TRIAL: NCT04146610
Title: A Phase Ia, Multicenter, Open and Dose-increasing Study of DP303c to Evaluate the Safety , Pharmacokinetics, Immunogenicity and Antitumor Activity of Subjects With HER2-Positive Advanced Solid Tumors
Brief Title: Study of DP303c Administered Intravenously to Subjects With HER2-Positive in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP303c201801
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dp303c (Experimental): Multiple dose grouping
  Interventions: Drug: an antibody drug conjugate

INTERVENTIONS:
Drug: an antibody drug conjugate — Multiple dose grouping
  Other Names: ADC

SUMMARY:
A phase Ia, multicenter, open and dose-increasing study of DP303c to evaluate the safety , pharmacokinetics, immunogenicity and antitumor activity of subjects with HER2-positive advanced solid tumors.

DETAILED DESCRIPTION:
Dose escalation study: Primary purpose: To investigate the safety and tolerability of DP303c in subjects with HER2-positive advanced solid tumors . Secondary purpose:1. To characterize the pharmacokinetics(PK) profile of DP303c;2. To assess the preliminary anti tumor activity of DP303c; 3. To characterize immunogenicity of DP303c.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent；
* Aged 18 to 75 years, both male and female;
* Patients with advanced solid tumors diagnosed by histology and / or cytology, confirmed to be HER2 positive by pathological examination, unable to accept or have no standard treatment, failure of standard treatment (disease progress or treatment without remission after treatment) or intolerable patients; HER2-positive is defined as IHC 2+ and ISH positive or IHC 3+； IHC scores of breast cancer and gastric cancer are based on their respective standards, while IHC scores of other cancers are based on the scoring standards of breast cancer；
* The ECOG performance status is 0 to 1,and the expected survival time is more than 3 months；
* Subjects must have laboratory values within the limits described below:

ANC ≥1.5 x 109/L Platelet count ≥100 x 109/L Hemoglobin ≥9 g/dL Serum creatinine within normal limits OR creatinine clearance ≥60 mL/minute Serum total bilirubin ≤1.5 x ULN (up to 3 x ULN in subjects with Gilbert's syndrome) AST (SGOT) and ALT (SGPT) ≤2.5 x ULN (OR ≤5 X ULN for subjects with liver metastases) PT/INR and APTT ≤1.5 x ULN

* According to the RECIST v1.1 standard, there must be a measurable lesion at the base line；
* WOCBP must have a negative pregnancy test prior to study entry；
* WOCBP and male subjects must agree to use adequate contraception from study entry through at least 12 weeks after the last dose of study drug (see Appendix 5)；
* A washout period is required for subjects who have recently received systemic antitumor therapy. The period prior to the subject's planned first dose of DP303c must be either at least 28 days or 5 half-lives, whichever is shorter. Antitumor therapy includes chemotherapy, immunotherapy, targeted therapy, endocrine therapy, radiotherapy (except local radiotherapy for pain relief, 14 days after treatment).

Exclusion Criteria:

* Pregnant or breastfeeding women；
* Refusal to use effective methods of contraception (see inclusion criteria for details)；
* Not recovered from AEs caused by previous drugs or radiotherapy (reference NCI CTCAE 5.0, ≤Grade 1 or at baseline), with the exception of alopecia；
* History of cardiac dysfunction with LVEF <40% while on trastuzumab therapy；
* Subjects with a history of allergy to any components(tratozumab analogues, MMAE, sodium citrate dihydrate, citrate monohydrate, polysorbitol 20 and sucrose, etc.) of DP303cand those who researchers consider to be more serious；
* A history of central nervous system (CNS) metastases or epilepsy, asymptomatic or stable, and not requiring treatment at least 4 weeks before study therapy began；
* Active lung infection or pneumonitis or a history of non-infectious interstitial lung disease；
* Requires supplemental oxygen；
* History of congestive heart failure, unstable angina pectoris, unstable atrial fibrillation, or cardiac arrhythmia. Subjects who have the following types of cardiac impairment at the time of enrollment:

New York Heart Association class III or IV heart disease Uncontrolled angina, congestive heart failure, or myocardial infarction within 6 months prior to enrolment An LVEF by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan <50% or below the lower limit of normal for the institution QT interval prolongation (>450 ms in males, >470 ms in females),QT interval correction (QTcF) was corrected by Fridericia formula

* In the first 90 daysof the study, Cumulative anthracycline dose ≥360 mg/m2 doxorubicin or equivalent；
* Peripheral neuropathy ≥Grade 2 or greater (NCI CTCAE v 5.0)；
* 12.Non-manageable electrolyte imbalances including hypokalemia, hypocalcemia, or hypomagnesemia (≥Grade 2 or greater based on NCI CTCAE v 5.0)；
* Any uncontrollable intercurrent illness, infection, or other conditions that could limit study compliance or interfere with assessments；
* Serologic status reflecting active hepatitis B or C infection；
* Subjects with immunodeficiency, including HIV positive；
* Patients were treated with CYP3A inhibitors within 14 days of the first dose (drugs that increased specific CYP substrate AUC ≥ 5 times, such as Mibefradil, verapamil, diltiazem, nefazodone, clarithromycin, Telithromycin, Troleandomycin, Erythromycin, fluconazole, itraconazole, ketoconazole, Posaconazole,VoriconazoleTablets，Elvitegravir，indinavir，lopinavir， Nelfinavir，Ritonavir，Saquinavir， Boceprevir，Incivo，telaprevir，Conivaptan，idelalisib) or strong CYP3A inducers (Avasimibe, phenobarbital, phenytoin, carbamazepine,Rifampicin, rifabutin,enzalutamide, mitotane, Hypericum perforatum )；
* Other serious or uncontrollable diseases or conditions that may affect the assessment of the primary endpoint or that the investigator considers to be at risk for participants participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Maximal Tolerance Dose (MTD) of Dp303c | The first treatment cycle 21 days
  The dose level in which >= 2 out of 6 patients have dose-limiting toxicity (DLT). The MTD is defined as the previous dose level.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of DP303c | approximately 2 years
  The pharmacokinetics(PK) profile of DP303c
Time of peak plasma concentration (Tmax) | approximately 2 years
  The pharmacokinetics(PK) profile of DP303c
Area under the plasma concentration time curve (AUC) of DP303c | approximately 2 years
  The pharmacokinetics(PK) profile of DP303c
Overall response rate (ORR) | approximately 2 years
  To preliminarily evaluate ORR in patients with advanced solid tumors.
Duration of Response (DoR) | approximately 2 years
  To preliminarily evaluate DoR in patients with advanced solid tumors.
Immunogenicity (anti-drug antibody ADA) | approximately 2 years
  Percentage of subjects producing detectable anti-drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Du Y, Meng Y, Liu X, Mu Y, Liu Y, Shi Y, Wang J, Zang A, Gu S, Liu T, Zhou H, Guo H, Xiang S, Zhang X, Wu S, Qi H, Li M, Hu X. First-in-human study of DP303c, a HER2-targeted antibody-drug conjugate in patients with HER2 positive solid tumors. NPJ Precis Oncol. 2024 Sep 12;8(1):200. doi: 10.1038/s41698-024-00687-7. PMID 39266619